CLINICAL TRIAL: NCT05050006
Title: A Phase 2, Open-label, Multicenter Study Evaluating the Safety and Efficacy of Autologous Tumor-infiltrating Lymphocytes (TILs) in Subjects With Advanced Melanoma (DELTA-1)
Brief Title: ITIL-168 in Advanced Melanoma
Acronym: DELTA-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Instil Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITIL-168-101; 2020-003862-37 (EudraCT Number)
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Advanced Cutaneous Melanoma
Keywords: ITIL-168; Cell Therapy; melanoma; Autologous cell therapy; Cellular Immunotherapy; TIL; Autologous Adoptive Cell Transfer; Immuno-oncology; IL-2; Autologous Adoptive Cell Therapy; Tumor Infiltrating Lymphocytes; T-cell therapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: All enrolled participants are assigned to be treated with a single dose of ITIL-168
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Patients who relapsed after or were refractory to at least 1 prior line of systemic therapy including a PD-1 inhibitor.
  Interventions: Biological: ITIL-168
- Cohort 2 (Experimental): Patients who were intolerant to a PD-1 inhibitor and have persistent disease after stopping PD-1 therapy.
  Interventions: Biological: ITIL-168
- Cohort 3 (Experimental): Patients who had a best response of stable disease despite being treated with at least 4 doses of a PD-1 inhibitor in the previous line of therapy.
  Interventions: Biological: ITIL-168

INTERVENTIONS:
Biological: ITIL-168 — ITIL-168 is a cell therapy product derived from a patient's own TILs. A tumor sample is removed from each patient to make a personalized ITIL-168 product. Once ITIL-168 has been made, the patient is treated with 5 days of lymphodepleting chemotherapy including cyclophosphamide and fludarabine, followed by a single infusion of ITIL-168, and up to 8 doses of IL-2.

SUMMARY:
DELTA-1 is a phase 2 clinical trial to evaluate the efficacy and safety of ITIL-168 in adult subjects with advanced melanoma who have previously been treated with a PD-1 inhibitor. ITIL-168 is a cell therapy derived from a patient's own tumor-infiltrating immune cells (lymphocytes; TILs).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed advanced (unresectable or metastatic) cutaneous melanoma.
* Cohort 1: Disease that is relapsed after or refractory to at least 1 prior line of systemic therapy that must include a PD-1 inhibitor and, if positive for proto- oncogene BRAF V600 activating mutation, targeted therapy.
* Cohort 2: Disease that is persistent after discontinuing PD-1 due to toxicity. Patients with a proto-oncogene BRAF V600 activating mutation must have progressed after targeted therapy.
* Cohort 3: Disease that is stable (SD) after at least 4 doses of a PD-1 inhibitor. Patients with a proto-oncogene BRAF V600 activating mutation must have progressed after targeted therapy.
* Medically suitable for surgical resection of tumor tissue
* Following tumor resection for TIL harvest, will have, at minimum, 1 remaining measurable lesion as identified by CT or MRI per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow and organ function

Key Exclusion Criteria:

* History of another primary malignancy within the previous 3 years
* Melanoma of uveal, acral, or mucosal origin
* Previously received an allogeneic stem cell transplant or organ allograft
* Previously received TIL or engineered cell therapy ( eg, CAR T-cell)
* Significant cardiac disease
* Stroke or transient ischemic attack within 12 months of enrollment
* History of significant central nervous system (CNS) disorder
* Symptomatic and/or untreated CNS metastases
* History of significant autoimmune disease within 2 years prior to enrollment
* Known history of severe, immediate hypersensitivity reaction attributed to cyclophosphamide, fludarabine, or IL-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 60 months
  Objective response rate (ORR), defined as the incidence of a complete response (CR) or a partial response (PR) per a modified Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria, as assessed by central review.

SECONDARY OUTCOMES:
Duration of Response | Up to 60 months
  For subjects who experience an objective response, duration of response (DOR) is defined as the time from their first objective response to disease progression or death.
Progression-free Survival | Up to 60 months
  Progression-free survival (PFS) is defined as the time from the ITIL-168 infusion date to the date of disease progression or death from any cause.
Overall Survival | Up to 60 months
  Overall survival (OS) is defined as the time from the ITIL-168 infusion date to the date of death from any cause.
ORR as determined by investigators | Up to 60 months
  ORR as determined by investigators is defined as the incidence of a CR or a PR per a modified RECIST v1.1, as determined by study investigators.
Frequency, duration, and severity of ITIL-168 treatment-emergent adverse events (AEs), serious AEs, and AEs of special interest | Up to 60 months
Disease Control Rate | Up to 60 months
  Disease control rate (DCR), defined as the incidence of CR, PR, or stable disease (SD) per a modified RECIST v1.1 criteria, as determined by central review.
Best Overall Response | Up to 60 months
Time to Response | Up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Instil Study Director, Study Director — Instil Bio, Inc.
Locations (22):
- United States (20):
  - University of California San Diego, Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC - Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Health - Westwood Cancer Care, Los Angeles, California
  - Stanford Cancer Institute, Stanford, California
  - University of Colorado - Anschutz Cancer Pavilion, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - The University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Rush University Cancer Center, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Cambridge University Hospital NHS Foundation Trust - Addenbrooke's Hospital, Cambridge, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No